CLINICAL TRIAL: NCT02885844
Title: Effects of Inverted Vision on Pointing and Grasping in Parabolic Flight
Acronym: SpaceInVision
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Collaborators: International Space University (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2014-A00813-44; NCT02517203 (obsolete NCT alias)
Record Dates: First submitted 2016-03-08; First posted 2016-09-01 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2016-05

CONDITIONS: Pointing Task; Gasping Task

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- INVERTED VISION (Experimental): inverted vision (upside down) using commercial off-the-shelf inverting prism goggles
  Interventions: Procedure: INVERTED VISION
- NORMAL VISION (Active Comparator): During normal vision trials, subject's field of view will be restricted by goggles without lenses (see below) in order to be equivalent to the inverted vision one.
  Interventions: Procedure: NORMAL VISON

INTERVENTIONS:
Procedure: INVERTED VISION — The tasks will be performed either with normal or inverted vision (upside down) using commercial off-the-shelf inverting prism goggles
  Arms: INVERTED VISION
Procedure: NORMAL VISON — subject's field of view will be restricted by goggles without lenses in order to be equivalent to the inverted vision one.
  Arms: NORMAL VISION

SUMMARY:
Parabolic flight is the only ground-based condition in which weightlessness (0G) can be created long enough for safely testing changes in human perception and behavior. In addition to the 0G period, parabolic flight generates equal duration periods of 1.8G, which present another unique opportunity to test the same responses to hypergravity and back to 1G.

Spatial orientation perception is a critical subsystem that is used by the central nervous system in the control of vehicles and other complex systems in a high-level integrative function. Evidence from space flight research demonstrates that spatial orientation is altered by the transitions in gravito-inertial force levels (Clément 2011; Clément & Reschke 2008), transitions corresponding to mission phases particularly critical for crew safety and mission success. Accurate perception of self-in-space motion and self-motion relative to other objects is critical for successful operations that involve motor control e.g. doing an extra-vehicule activity or piloting the spacecraft. To date, there is only limited operational evidence that these alterations cause functional impacts on mission-critical operations and control capabilities. Immediately after space flight, most crewmembers have reported some degree of disorientation/perceptual illusion, often accompanied by nausea (or other symptoms of motion sickness), and frequently manifested by lack of coordination, particularly during locomotion The hypothesis is that alteration in sensorimotor performance induced by inverted vision is gravity depend: maximum alteration during hypergravity, intermediary alteration during normal gravity, minimal alteration during weightlessness.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be staff member of the team or of other teams participating in the parabolic flight campaign
* Healthy volunteers (men or women)
* Aged from 21 to 65
* Affiliated to a Social Security system and, for non-French resident, holding a European Health Insurance Card (EHIC)
* Who accepted to take part in the study
* Who have given their written stated consent
* Who has passed a medical examination similar to a standard aviation medical examination for private pilot aptitude (JAR FCL3 Class 2 medical examination). There will be no additional test performed for subject selection.

Exclusion Criteria:

* Person who took part in a previous biomedical research protocol, of which exclusion period is not terminated
* Person with medical history of oculomotor disorders
* Person with medical history of vestibular disorders
* Pregnant women

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2014-09; Primary Completion 2017-09 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Response time | During flight
  the time between when the target or shape appears and the subject lifts their finger off of the screen

SECONDARY OUTCOMES:
Task duration | During flight
  Only for the grasping task - the time between when the subject lifts their finger from the screen after having seen the shape, grasps the shape and touches the screen again. This will also be measured for the time between when the subject touches the screen, places the shape in the correct form fitter and touches the screen again
Accuracy | During flight
  Only for the pointing task - the measured Euclidian distance from the target center to the coordinates of where the subject touched the screen.

CONTACTS AND LOCATIONS:
Overall Officials: Clément GC Gilles, Study Director — International Space University
Locations (1):
- CHU Caen, Caen, France

IPD SHARING:
Plan to Share IPD: No